CLINICAL TRIAL: NCT06285591
Title: Lactobacillus Reuteri Alleviates Oral Mucositis in Patients Undergoing Radiotherapy for Malignant Head and Neck Tumors: A Randomized Controlled Trial
Brief Title: Lactobacillus Reuteri Alleviates Oral Mucositis in Patients Undergoing Radiotherapy for Malignant Head and Neck Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-1801
Record Dates: First submitted 2024-02-06; First posted 2024-02-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Malignant Tumors
Keywords: Head and Neck Malignant Tumors; Radiation-induced oral mucositis; Lactobacillus reuteri
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Placebo-containing tablets
  Interventions: Drug: Placebo-containing tablets; Radiation: Radiotherapy
- Experimental group (Experimental): Lactobacillus reuteri tablets
  Interventions: Drug: Lactobacillus reuteri Tablets; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Lactobacillus reuteri Tablets — Lactobacillus reuteri lozenges (NOW Foods, Sweden) contained 2×10^8 CFU viable cells of Lactobacillus reuteri as the active ingredient.
  Arms: Experimental group
Drug: Placebo-containing tablets — The placebo lozenges shared the same formulation as the L. reuteri lozenges but without the probiotic, whose appearance, taste, and color were identical to those of the Lactobacillus reuteri lozenges.
  Arms: Control group
Radiation: Radiotherapy — One of the inclusion criteria for the study was that patients with malignant tumors of the head and neck (including nasopharyngeal carcinoma) needed to receive either radiotherapy alone or simultaneous radiotherapy and chemotherapy.

SUMMARY:
To evaluate the efficacy and safety of Lactobacillus reuteri for prevention and treatment of oral mucositis in patients undergoing radiotherapy for malignant head and neck tumors.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the efficacy and safety of Lactobacillus reuteri in reducing the incidence, duration, and severity of severe oral mucositis (SOM). The main questions it aims to answer are whether Lactobacillus reuteri can effectively prevent and treat radiation-induced oral mucositis and whether it will cause adverse events in patients undergoing radiotherapy.

Participants will be instructed to suck a Lactobacillus reuteri or placebo lozenge twice daily from the beginning to the end of RT. After using the lozenges, the patients should avoid eating, drinking and conducting any oral hygiene activities for at least 1 hour.

Researchers will compare Lactobacillus reuteri group and placebo group to see if oral probiotic are beneficial in preventing and treating oral mucositis in patients undergoing radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients pathologically diagnosed with non-metastatic head and neck malignant tumors;
2. Aged 18-80 years;
3. Eastern Cooperative Oncology Group performance status of ≤2;
4. Receiving definitive RT or postoperative adjuvant RT at a dose of 60-72Gy with/without concurrent chemotherapy;
5. Sign informed consent.

Exclusion Criteria:

1. Patients with known allergy to probiotic or severe allergic constitution;
2. Use of antibiotics, antifungal drugs, or antimicrobial mouthwash within 1 month of the study;
3. Poor oral hygiene and/or severe periodontal diseases;
4. History of head and neck radiotherapy;
5. Deemed unsuitable for the study by the investigators (concomitant with any other severe diseases).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
The incidence of severe oral mucositis (SOM) (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Oral mucositis is assessed by trained radiotherapists according to World Health Organization (WHO) oral toxicity Scale.The WHO Oral Toxicity Scale categorizes oral mucositis into grades 0-4, with the higher the grade the more severe the patient's oral mucositis. Grade 0 means that the oral mucosa is normal and the patient has no symptoms or signs; grade 1 means that the mucosa is erythematous with or without pain and does not interfere with eating; grade 2 means that the mucosa is erythematous and ulcerated, but still able to eat solid food; grade 3 means that the mucosa is severely ulcerated with extensive erythema and unable to eat solid food; and grade 4 means that the ulcers of the mucosa are fused together into a sheet, and their severity is so severe that it is not possible to eat.

SECONDARY OUTCOMES:
The time to onset of severe oral mucositis (SOM) (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Time from the first day of radiotherapy to the first determination of SOM.
The duration of severe oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  The first determination of SOM to the first instance of non-severe OM (WHO grade <3), without a subsequent instance of SOM.
The incidence of oral mucositis (OM) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Oral mucositis is assessed by trained physicians according to World Health Organization (WHO) oral toxicity Scale.
The time to onset of any-grade oral mucositis (OM) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  Time from the first day of radiotherapy to the first determination of OM.
The duration of any-grade oral mucositis (OM) | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks and 14.5 weeks.
  The first determination of OM to the first instance of non-OM, without a subsequent instance of OM.

OTHER OUTCOMES:
Quality of life as sssessed by the EORTC QLQ-C30 and QLQ-H&N35 Questionnaires | 1 week before radiotherapy ; at the middle of radiotherapy (usually 3 weeks after the start of radiotherapy) ; at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks) ; and 1, 2, 3 months after the end of radiotherapy.
  European Organization for Research and Treatment of Cancer (EORTC) Quality-of-life Questionnaire Core 30 (EORTC QLQ-C30) and Head and Neck Cancer Module (EORTC QLQ-H&N35).
Mouth and throat soreness score | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  Patients report two scores via the Oral Mucositis Weekly Questionnaire (OMWQ): (1) the severity of mouth and throat soreness (MTS) and (2) the degree of its impact on oral activities (including swallowing, drinking, eating, talking, and sleeping). Both items use a Likert scale from 1 to 5, with higher scores indicating more severe symptoms or greater functional impairment.
Hyposalivation | 1 week before radiotherapy ; at the middle of radiotherapy (usually 3 weeks after the start of radiotherapy) ; at the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks); and 1, 3 months after the end of radiotherapy.
  Hyposalivation was graded per CTCAE v5.0 (Grade 1-4), with higher grades indicating worse symptoms.
Gustatory function | 1 week before radiotherapy ; at the middle of radiotherapy (usually 3 weeks after the start of radiotherapy) ; at the end of radiotherapy（the last radiation dose received, usually 6 or 6.5 weeks） ; and 1, 3 months after the end of radiotherapy.
  Taste strips test.
Change in weight | The time period is the period from the start of radiotherapy to the completion of radiotherapy. The evaluation period is approximately 6 weeks and 6.5 weeks.
  The change in patient's body weight measured at baseline (pre-radiotherapy) and at the end of radiotherapy.
The number of patients receiving parenteral nutrition | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  This outcome records the number of patients who receive parenteral nutrition from the start to the completion of radiotherapy.
The number of patients receiving analgesics | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  This outcome records the number of patients who receive analgesics from the start to the completion of radiotherapy.
Radiotherapy interruption rate | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  The number of patients who missed five or more consecutive radiations and the reasons for this are recorded during radiotherapy.
Adverse events | From the first day of radiotherapy to the day of the last radiation dose received, usually 6 or 6.5 weeks.
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version
The composition and dynamics of salivary microbiota | 1 week before radiotherapy, the middle of radiotherapy (usually 3 weeks after the start of radiotherapy), and the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks).
  Unstimulated whole saliva samples will be collected via spitting method at three time points: baseline, mid-term radiotherapy (the week corresponding to 50% completion of the planned radiation fractions), and the end of radiotherapy (the final week of RT). 16S rRNA gene sequencing will be performed to assess alterations in the oral microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No